CLINICAL TRIAL: NCT06808828
Title: Occupational Therapy for Adults Who Have Experienced Intimate Partner Violence
Brief Title: Occupational Therapy for Adults Who Have Experienced Intimate Partner Violence (IPV)
Acronym: IPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5240501
Record Dates: First submitted 2025-01-25; First posted 2025-02-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Domestic Violence
Keywords: domestic violence; intimate partner violence; occupational therapy
MeSH Terms: interventions — Health; Coping Skills

STUDY DESIGN:
Intervention Model Description: Participants will attend a 90-minute session twice a week sessions per week for four weeks. During the session, participants will receive education on resilience and developing healthy lifestyles. Participants will be assessed at baseline with a pre-test and post-intervention with a post-test. In addition, participants will complete the occupational therapy lifestyle medicine check-in at each session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health and coping skills (Experimental): Subjects will complete an 8-item occupational therapy lifestyle medicine checklist at each session. The subjects will participate in eight sessions receiving education on health topics of sleep hygiene, physical activity, healthy cooking, self-management, coping skills, self-esteem, mindfulness, and goal setting.
  Interventions: Behavioral: Health and coping skills

INTERVENTIONS:
Behavioral: Health and coping skills — An occupational therapist and occupational therapy graduate capstone student will lead in-person sessions. Subjects will participate in an occupational therapy program that meets 2x/week x 4 weeks for eight sessions. Topics will include sleep hygiene, physical activity, healthy cooking, self-management, coping skills, self-esteem, mindfulness, and goal setting. Subjects will receive education as well as actively engage in activities related to the topic. Subjects will be provided with a personal journal to complete homework involving reflections on the topics discussed in the sessions.

SUMMARY:
The purpose of this graduate student research study is to understand the effectiveness of an occupational therapy program in a domestic violence shelter. It is expected that participation will last about 6 weeks. Subjects will complete pretests involving lifestyle assessments and a coping scale and then participate in 8 occupational therapy sessions during the 4 weeks of program implementation. The occupational therapy sessions will last approximately 90 minutes. After the program is completed, subjects will complete the posttests.

Procedures and Activities. You will be asked to:

Complete a series of questionnaires about your health, well-being, and daily activities.

Participate in 8 OT sessions that may include activities such as journaling, positive self-talk, coping skills methods, and grounding exercises.

Complete the posttests.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 years of age or older receiving services from a domestic violence organization

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in Healthy Lifestyle | Change between baseline assessment at initial enrollment and completion of Session 8 at 8 weeks post-enrollment.
  This is a composite measurement, utilizing the Occupational Therapy Lifestyle Medicine Checklist (OTLM) to assess improvement in the following categories: Healthy eating; Physical Activity; Stress Management; Social Connections; Sleep; Work/School (that's too vague to measure), Leisure and Hobbies; Avoiding Risky Substances. Participants will complete this checklist at baseline, prior to the first intervention and after the final eight intervention is completed. Each category will have a range (1-10), which will indicate how the participant has responded overall to the intervention. An overall increase of >15 points in the combined categories will indicate significant improvement. An overall decrease of any number of points will indicate non-significant improvement.
Improvement in Quality of Life | Change between the baseline assessment and post-test at study completion, up to 9 weeks post-enrollment
  This is a compositive measure utilizing the 36-Item Short Form Health Survey Questionnaire. Quality of life involves several areas. The 36-item Short Form is a self-reported measure that consists of thirty-six questions covering eight domains of health. Categories include (1) limitations in physical activities, (2) limitations in social activities, (3) limitations in usual role activities because of physical health problems, (4) bodily pain, (5) general mental health, (6) limitations in usual role activities because of emotional problems, (7) vitality, and (8) general health perceptions. Subjects may receive a score ranging from 0-100. Higher scores indicate more favorable health.
Improvement in Coping Skills | Change between the baseline assessment and post-test at study completion, up to 9 weeks post-enrollment.
  This is a composite measure that will utilize the Coping Scale Questionnaire. This 13-item questionnaire gathers information on how the subject copes. Categories include anger management, endurance, well-being, and posttraumatic growth. Higher scores indicate higher levels of coping.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Javaherian, OTD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No